CLINICAL TRIAL: NCT07403500
Title: Evaluation of the Short-term Effectiveness of Spinal Manipulation to Treat Acute and Subacute Low Back Pain. An Open-label Randomized Controlled Multicenter Trial.
Brief Title: Evaluation of the Short-term Effectiveness of Spinal Manipulation to Treat Acute and Subacute Low Back Pain.
Acronym: MeLoPe
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESPIR/2022/AD-01
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Back Pain Lower Back Chronic
Keywords: Back; Pain; Chronic; Spinal manipulation
MeSH Terms: conditions — Pain; Bronchiolitis Obliterans Syndrome | interventions — Physical Therapy Modalities

STUDY DESIGN:
Masking Description: As it is not possible to conduct this trial blinded or even with a blinded evaluator, in order to limit the detrimental effect of subjectivity, the word "placebo" will not be mentioned in the information given to patients (verbal information provided by investigators and written information sheet) and the meaning of the hypothesis will not be mentioned either. The aim will be to compare two types of manipulation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPINE MANIPULATION (SM) (Experimental): The physician determines the level(s) with segmental dysfunction(s), checks the conditions for performing MV (free directions of trunk movement, absence of red flags), which consists of a dynamic push at high speed and low amplitude, a lateral rotation push in flexion performed on one or more vertebral segments where minor intervertebral disturbances are located (patient lying on their side). The rationale behind this approach is to treat minor intervertebral disturbances causing lumbar pain by activating a reflex mechanism that allows muscle relaxation.
  Interventions: Other: Spinal or peripheral manipulation of the lower back to treat lower back pain
- PERIPHERAL MANIPULATION (PM) (Active Comparator): The doctor determines the level(s) with segmental dysfunction(s), then performs peripheral treatment using osteopathic techniques, offering comprehensive treatment for the patient. Mobilization and palpation are localized in the lower limbs (knee and ankle), the abdomen with massage of the psoas muscles, the upper limbs (shoulder and elbow), and the cervical spine with high-amplitude, low-speed mobilization without thrusting. The rationale behind this approach is the treatment of an overall imbalance causing back pain and requiring rebalancing.
  Interventions: Other: Spinal or peripheral manipulation of the lower back to treat lower back pain

INTERVENTIONS:
Other: Spinal or peripheral manipulation of the lower back to treat lower back pain — The patient will receive treatment for lower back pain (spinal or peripheral manipulation) according to their assignment group.
  Other Names: Physiotherapy

SUMMARY:
Low back pain is the second most common reason for medical consultation in France and affects 60 to 80% of the working population. Patients with acute episodes of non-specific low back pain recover within 6 to 8 weeks, but recurrence is common and 7 to 10% of patients will experience persistent pain and disability for more than 3 months. Given their low efficacy and the risks associated with nonsteroidal anti-inflammatory drugs or opioids (nearly 60% of all opioids prescribed in the United States), the scientific literature does not support the use of pharmacological treatments. The international recommendations strongly suggest using non-pharmacological therapies, including physical exercise, rehabilitation, and spinal manipulation.Spinal manipulation (SM) is a common choice of therapy in primary care. In the patient's imagination "getting manipulated when in pain leads to heavy use of these manual therapies in a medical (manual medicine and medical osteopathy) or non-medical setting (manual therapy, osteopathy, and chiropractic). However, the evidence of effectiveness is weak in the chronic phase (only in the short term) and contradictory for the acute or subacute phases of low back pain. Pain and function are improved at 6 weeks, but the results are not clinically relevant. There is a lack of evidence regarding efficacy because the trials on spinal manipulations are of poor quality. A meta-analysis has recently reported that SMs are associated with a very limited risk of harm, making them a reasonable treatment option. Therefore, it seems necessary to demonstrate the specific effect of MVs in order to justify their use in primary care, support their wider use around the world, and reinforce recommendations for non-pharmacological treatment of low back pain.

DETAILED DESCRIPTION:
Low back pain is a common musculoskeletal condition that affects 60 to 80% of the working population at least once in their lifetime. Patients with acute episodes of non-specific low back pain recover within 6 to 8 weeks, but recurrence is common and 7 to 10% of them will experience persistent pain and disability for more than 3 months. It is the second most common reason for medical consultation in France.

The scientific literature does not support the use of pharmacological treatments given their low efficacy and the risks associated with prescribing nonsteroidal anti-inflammatory drugs or opioids (which account for nearly 60% of all opioids prescribed in the United States). It is therefore easy to understand why the international recommendations strongly suggest using non-pharmacological therapies, including physical exercise, rehabilitation, and spinal manipulation.

Spinal manipulation (SM) is a very common therapy of choice in primary care, enjoying popularity beiliefs rooted in the patient's imagination ("getting manipulated when you're in pain"), leading to heavy use of these manual therapies in a medical (manual medicine and medical osteopathy) or non-medical setting (manual therapy, osteopathy, and chiropractic). However, evidence of effectiveness is considered weak in the chronic phase (only in the short term) and contradictory for the acute or subacute phases of low back pain. Pain and function are improved at 6 weeks, but the results are not clinically relevant. The main reason for this lack of evidence is that efficacy trials concerning spinal manipulations are, at best, of poor quality for a number of reasons: SMs are very often combined with other strategies (exercises, medication, rehabilitation, etc.), which limits the assessment of a specific effect; manual therapies are very diverse, limiting comparability; the time required to assess the effects is often long (more than 4 weeks), comparable to the usual time required for pain to resolve; comparative trials are of low power, limiting the ability to demonstrate a difference; The use of a placebo comparator to test the effect of MV is not trivial and must be carefully defined, particularly for physicians who do not consider placebo to be an alternative in standard care. As far as we know, there has only been one RTC against placebo, the results of which were negative (n=240).

A meta-analysis has recently reported that SMs are associated with a very limited risk of harm, making them a reasonable treatment option. Therefore, it seems necessary to demonstrate the specific effect of MVs in order to justify their use in primary care, support their wider use around the world, and reinforce recommendations for non-pharmacological treatment of low back pain.

The hypothesis is that patients receiving spinal manipulations will experience greater pain relief in the short term (7 to 10 days after treatment) than patients receiving peripheral manipulations.

Patients in the experimental group (spinal manipulation) should also show improvement in their pain in the medium term, their functional abilities, their physical and work avoidance scores, catastrophizing, and the occurrence of lumbar flare-ups up to three months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking treatment for low back pain present for less than 3 months, with an average intensity greater than 50 on a visual analog scale of 0-100 in the previous 48 hours.
* Patients able to complete online questionnaires.
* Patients who have given their free and informed consent.
* Patients who are affiliated with or beneficiaries of a health insurance plan.

Exclusion Criteria:

* Patients with a history of back surgery, undergoing corticosteroid or morphine treatment, with acute or chronic inflammatory diseases, with psychiatric illness, or with low back pain lasting more than 3 months.
* Patients who have already undergone spinal manipulation for low back pain with the investigator.
* Patients participating or having participated in a therapeutic or drug study in the 3 months prior to their inclusion in this protocol.
* Patients in a period of exclusion determined by another study.
* Patients under legal protection, guardianship, or conservatorship.
* Patients unable to give their consent.
* Patients for whom it is impossible to provide informed consent.
* Pregnant or breastfeeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Short-term effectiveness (7 to 10 days) of spinal manipulation (SM) on pain over the last 24/48 hours in acute and subacute low back pain : experimental group | Day 0
  Pain assessment using a visual analog scale of 0-100 over the last 24/48 hours
Short-term effectiveness (7 to 10 days) of spinal manipulation (SM) on pain over the last 24/48 hours in acute and subacute low back pain : experimental group | Day 7
  Pain assessment using a visual analog scale of 0-100 over the last 24/48 hours
Short-term effectiveness (7 to 10 days) of spinal manipulation (SM) on pain over the last 24/48 hours in acute and subacute low back pain : experimental group | Day 10
  Pain assessment using a visual analog scale of 0-100 over the last 24/48 hours
Short-term effectiveness (7 to 10 days) of peripheral manipulation (PM) on pain over the last 24/48 hours in acute and subacute low back pain : control group | Day 0
  Pain assessment using a visual analog scale of 0-100 over the last 24/48 hours
Short-term effectiveness (7 to 10 days) of peripheral manipulation (PM) on pain over the last 24/48 hours in acute and subacute low back pain : control group | Day 7
  Pain assessment using a visual analog scale of 0-100 over the last 24/48 hours
Short-term effectiveness (7 to 10 days) of peripheral manipulation (PM) on pain over the last 24/48 hours in acute and subacute low back pain : control group | Day 10
  Pain assessment using a visual analog scale of 0-100 over the last 24/48 hours

SECONDARY OUTCOMES:
Evolution of lower back pain and lower limb pain (above the knee) in the experimental group (SM) | Day 1 to 2
  Measurement of pain in the back and lower limbs at rest and during activities over the last 24/48 hours at 7/10 days and 3 weeks, then at 1 and 3 months using the visual analog pain scale (0-100).
Evolution of lower back pain and lower limb pain (above the knee) in the control group (PM) | Day 1 to 2
  Measurement of pain in the back and lower limbs at rest and during activities over the last 24/48 hours at 7/10 days and 3 weeks, then at 1 and 3 months using the visual analog pain scale (0-100).
Evolution of lower back pain and lower limb pain (above the knee) in the experimental group (SM) | Day 7 - 10
  Measurement of pain in the back and lower limbs at rest and during activities over the last 24/48 hours at 7/10 days and 3 weeks, then at 1 and 3 months using the visual analog pain scale (0-100).
Evolution of lower back pain and lower limb pain (above the knee) in the control group (PM) | Day 7 - 10
  Measurement of pain in the back and lower limbs at rest and during activities over the last 24/48 hours at 7/10 days and 3 weeks, then at 1 and 3 months using the visual analog pain scale (0-100).
Evolution of lower back pain and lower limb pain (above the knee) in the experimental group (SM) | Week 3
  Measurement of pain in the back and lower limbs at rest and during activities over the last 24/48 hours at 7/10 days and 3 weeks, then at 1 and 3 months using the visual analog pain scale (0-100).
Evolution of lower back pain and lower limb pain (above the knee) in the control group (PM) | Week 3
  Measurement of pain in the back and lower limbs at rest and during activities over the last 24/48 hours at 7/10 days and 3 weeks, then at 1 and 3 months using the visual analog pain scale (0-100).
Evolution of lower back pain and lower limb pain (above the knee) in the experimental group (SM) | Month 1
  Measurement of pain in the back and lower limbs at rest and during activities over the last 24/48 hours at 7/10 days and 3 weeks, then at 1 and 3 months using the visual analog pain scale (0-100).
Evolution of lower back pain and lower limb pain (above the knee) in the control group group (PM) | Month 1
  Measurement of pain in the back and lower limbs at rest and during activities over the last 24/48 hours at 7/10 days and 3 weeks, then at 1 and 3 months using the visual analog pain scale (0-100).
Evolution of lower back pain and lower limb pain (above the knee) in the experimental group (SM) | Month 3
  Measurement of pain in the back and lower limbs at rest and during activities over the last 24/48 hours at 7/10 days and 3 weeks, then at 1 and 3 months using the visual analog pain scale (0-100).
Evolution of lower back pain and lower limb pain (above the knee) in the control group (PM) | Month 3
  Measurement of pain in the back and lower limbs at rest and during activities over the last 24/48 hours at 7/10 days and 3 weeks, then at 1 and 3 months using the visual analog pain scale (0-100).
Changes in movement avoidance due to pain in the experimental group (SM) | Day 0
  Measured according to the Fear Avoidance Beliefs Questionnaire (FABQ) score for physical avoidance and work avoidance. The FABQ is a patient reported questionnaire which specifically focuses on how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability. The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24). The questionnaire takes approximately 10 minutes to complete.
Changes in movement avoidance due to pain in the experimental group (SM) | Day 7 to 10
  Measured according to the Fear Avoidance Beliefs Questionnaire (FABQ) score for physical avoidance and work avoidance. The FABQ is a patient reported questionnaire which specifically focuses on how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability. The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24). The questionnaire takes approximately 10 minutes to complete.
Changes in movement avoidance due to pain in the experimental group (SM) | Month 1
  Measured according to the Fear Avoidance Beliefs Questionnaire (FABQ) score for physical avoidance and work avoidance. The FABQ is a patient reported questionnaire which specifically focuses on how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability. The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24). The questionnaire takes approximately 10 minutes to complete.
Changes in movement avoidance due to pain in the experimental group (SM) | Month 3
  Measured according to the Fear Avoidance Beliefs Questionnaire (FABQ) score for physical avoidance and work avoidance. The FABQ is a patient reported questionnaire which specifically focuses on how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability. The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24). The questionnaire takes approximately 10 minutes to complete.
Changes in movement avoidance due to pain in the control group (PM) | Day 0
  Measured according to the Fear Avoidance Beliefs Questionnaire (FABQ) score for physical avoidance and work avoidance. The FABQ is a patient reported questionnaire which specifically focuses on how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability. The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24). The questionnaire takes approximately 10 minutes to complete.
Changes in movement avoidance due to pain in the control group (PM) | Day 7 to 10
  Measured according to the Fear Avoidance Beliefs Questionnaire (FABQ) score for physical avoidance and work avoidance. The FABQ is a patient reported questionnaire which specifically focuses on how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability. The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24). The questionnaire takes approximately 10 minutes to complete.
Changes in movement avoidance due to pain in the control group (PM) | Month 1
  Measured according to the Fear Avoidance Beliefs Questionnaire (FABQ) score for physical avoidance and work avoidance. The FABQ is a patient reported questionnaire which specifically focuses on how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability. The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24). The questionnaire takes approximately 10 minutes to complete.
Changes in movement avoidance due to pain in the control group (PM) | Month 3
  Measured according to the Fear Avoidance Beliefs Questionnaire (FABQ) score for physical avoidance and work avoidance. The FABQ is a patient reported questionnaire which specifically focuses on how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability. The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24). The questionnaire takes approximately 10 minutes to complete.
Catastrophizing in the experimental group (SM) | Day 0
  Catastrophizing will be measured using the PCS (Pain Catastrophizing Scale). The PCS is a self-assessment questionnaire to examine catastrophizing in clinical and nonclinical populations. The PCS consists of 13 statements containing a number of thoughts and feelings one may experience when having pain. The items are divided into the categories of rumination, magnification and helplessness, with each item scored on a 5-point scale.Using a 5-point Likert scale, from 0 (not at all) to 4 (always), people are asked to rate how often they experience the mentioned thoughts and feelings when they are in pain. Along with three subscale scores evaluating rumination, magnification, and helplessness, the overall score has a range of 0-52. Subscale Scores: Rumination: Items 8,9,10,11 Magnification: Items 6,7,13 Helplessness: Items 1,2,3,4,5,12. Higher scores indicate a greater degree of pain catastrophizing. A total score of >30 represents a clinically significant level of pain catastrophization.
Catastrophizing in the experimental group (SM) | Day 7 to 10
  Catastrophizing will be measured using the PCS (Pain Catastrophizing Scale). The PCS is a self-assessment questionnaire to examine catastrophizing in clinical and nonclinical populations. The PCS consists of 13 statements containing a number of thoughts and feelings one may experience when having pain. The items are divided into the categories of rumination, magnification and helplessness, with each item scored on a 5-point scale.Using a 5-point Likert scale, from 0 (not at all) to 4 (always), people are asked to rate how often they experience the mentioned thoughts and feelings when they are in pain. Along with three subscale scores evaluating rumination, magnification, and helplessness, the overall score has a range of 0-52. Subscale Scores: Rumination: Items 8,9,10,11 Magnification: Items 6,7,13 Helplessness: Items 1,2,3,4,5,12. Higher scores indicate a greater degree of pain catastrophizing. A total score of >30 represents a clinically significant level of pain catastrophization.
Catastrophizing in the experimental group (SM) | Month 1
  Catastrophizing will be measured using the PCS (Pain Catastrophizing Scale). The PCS is a self-assessment questionnaire to examine catastrophizing in clinical and nonclinical populations. The PCS consists of 13 statements containing a number of thoughts and feelings one may experience when having pain. The items are divided into the categories of rumination, magnification and helplessness, with each item scored on a 5-point scale.Using a 5-point Likert scale, from 0 (not at all) to 4 (always), people are asked to rate how often they experience the mentioned thoughts and feelings when they are in pain. Along with three subscale scores evaluating rumination, magnification, and helplessness, the overall score has a range of 0-52. Subscale Scores: Rumination: Items 8,9,10,11 Magnification: Items 6,7,13 Helplessness: Items 1,2,3,4,5,12. Higher scores indicate a greater degree of pain catastrophizing. A total score of >30 represents a clinically significant level of pain catastrophization.
Catastrophizing in the experimental group (SM) | Month 3
  Catastrophizing will be measured using the PCS (Pain Catastrophizing Scale). The PCS is a self-assessment questionnaire to examine catastrophizing in clinical and nonclinical populations. The PCS consists of 13 statements containing a number of thoughts and feelings one may experience when having pain. The items are divided into the categories of rumination, magnification and helplessness, with each item scored on a 5-point scale.Using a 5-point Likert scale, from 0 (not at all) to 4 (always), people are asked to rate how often they experience the mentioned thoughts and feelings when they are in pain. Along with three subscale scores evaluating rumination, magnification, and helplessness, the overall score has a range of 0-52. Subscale Scores: Rumination: Items 8,9,10,11 Magnification: Items 6,7,13 Helplessness: Items 1,2,3,4,5,12. Higher scores indicate a greater degree of pain catastrophizing. A total score of >30 represents a clinically significant level of pain catastrophization.
Catastrophizing in the control group (PM) | Day 0
  Catastrophizing will be measured using the PCS (Pain Catastrophizing Scale). The PCS is a self-assessment questionnaire to examine catastrophizing in clinical and nonclinical populations. The PCS consists of 13 statements containing a number of thoughts and feelings one may experience when having pain. The items are divided into the categories of rumination, magnification and helplessness, with each item scored on a 5-point scale.Using a 5-point Likert scale, from 0 (not at all) to 4 (always), people are asked to rate how often they experience the mentioned thoughts and feelings when they are in pain. Along with three subscale scores evaluating rumination, magnification, and helplessness, the overall score has a range of 0-52. Subscale Scores: Rumination: Items 8,9,10,11 Magnification: Items 6,7,13 Helplessness: Items 1,2,3,4,5,12. Higher scores indicate a greater degree of pain catastrophizing. A total score of >30 represents a clinically significant level of pain catastrophization.
Catastrophizing in the control group (PM) | Day 7 to 10
  Catastrophizing will be measured using the PCS (Pain Catastrophizing Scale). The PCS is a self-assessment questionnaire to examine catastrophizing in clinical and nonclinical populations. The PCS consists of 13 statements containing a number of thoughts and feelings one may experience when having pain. The items are divided into the categories of rumination, magnification and helplessness, with each item scored on a 5-point scale.Using a 5-point Likert scale, from 0 (not at all) to 4 (always), people are asked to rate how often they experience the mentioned thoughts and feelings when they are in pain. Along with three subscale scores evaluating rumination, magnification, and helplessness, the overall score has a range of 0-52. Subscale Scores: Rumination: Items 8,9,10,11 Magnification: Items 6,7,13 Helplessness: Items 1,2,3,4,5,12. Higher scores indicate a greater degree of pain catastrophizing. A total score of >30 represents a clinically significant level of pain catastrophization.
Catastrophizing in the control group (PM) | Month 1
  Catastrophizing will be measured using the PCS (Pain Catastrophizing Scale). The PCS is a self-assessment questionnaire to examine catastrophizing in clinical and nonclinical populations. The PCS consists of 13 statements containing a number of thoughts and feelings one may experience when having pain. The items are divided into the categories of rumination, magnification and helplessness, with each item scored on a 5-point scale.Using a 5-point Likert scale, from 0 (not at all) to 4 (always), people are asked to rate how often they experience the mentioned thoughts and feelings when they are in pain. Along with three subscale scores evaluating rumination, magnification, and helplessness, the overall score has a range of 0-52. Subscale Scores: Rumination: Items 8,9,10,11 Magnification: Items 6,7,13 Helplessness: Items 1,2,3,4,5,12. Higher scores indicate a greater degree of pain catastrophizing. A total score of >30 represents a clinically significant level of pain catastrophization.
Catastrophizing in the control group (PM) | Month 3
  Catastrophizing will be measured using the PCS (Pain Catastrophizing Scale). The PCS is a self-assessment questionnaire to examine catastrophizing in clinical and nonclinical populations. The PCS consists of 13 statements containing a number of thoughts and feelings one may experience when having pain. The items are divided into the categories of rumination, magnification and helplessness, with each item scored on a 5-point scale.Using a 5-point Likert scale, from 0 (not at all) to 4 (always), people are asked to rate how often they experience the mentioned thoughts and feelings when they are in pain. Along with three subscale scores evaluating rumination, magnification, and helplessness, the overall score has a range of 0-52. Subscale Scores: Rumination: Items 8,9,10,11 Magnification: Items 6,7,13 Helplessness: Items 1,2,3,4,5,12. Higher scores indicate a greater degree of pain catastrophizing. A total score of >30 represents a clinically significant level of pain catastrophization.
Occurrence and frequency of lumbar flare-ups in the 3 months following manipulation in the experimental group (SM) | Month 1
  The numbar of flare-ups, defined as episodes of low back pain greater than 50 out of 100 on the visual analog scale lasting more than 24 hours will be recorded. yes/no and if so, how many? Data collection via an online application made available to the patient.
Occurrence and frequency of lumbar flare-ups in the 3 months following manipulation in the experimental group (SM) | Month 3
  The numbar of flare-ups, defined as episodes of low back pain greater than 50 out of 100 on the visual analog scale lasting more than 24 hours will be recorded. yes/no and if so, how many? Data collection via an online application made available to the patient.
Occurrence and frequency of lumbar flare-ups in the 3 months following manipulation in the control group (PM) | Month 1
  The numbar of flare-ups, defined as episodes of low back pain greater than 50 out of 100 on the visual analog scale lasting more than 24 hours will be recorded. yes/no and if so, how many? Data collection via an online application made available to the patient.
Occurrence and frequency of lumbar flare-ups in the 3 months following manipulation in the control group (PM) | Month 3
  The numbar of flare-ups, defined as episodes of low back pain greater than 50 out of 100 on the visual analog scale lasting more than 24 hours will be recorded. yes/no and if so, how many? Data collection via an online application made available to the patient.
Functional disability in the experimental group (SM) | Day 0
  Functional disability will be measured according to the Roland Morris Disability Questionnaire (RMDQ). The RMDQ is scored by adding up the number of items checked by the patient. The score can therefore range from 0 to 24. The original version of the Roland Morris Disability Questionnaire was published by Roland and Morris in 1983. A review of articles on the questionnaire was published in 2000 (Roland & Fairbank 2000). It comprises 24 items and measures the functional disability of patients with low back pain. This self-administered questionnaire is quick, easy to use, reliable, valid, and sensitive to changes in clinical status, suggesting that its use could be generalized in contexts ranging from epidemiological or clinical research to the individual assessment of patients with low back pain in everyday clinical practice. The questionnaire takes approximately 5 minutes to complete.
Functional disability in the experimental group (SM) | Month 1
  Functional disability will be measured according to the Roland Morris Disability Questionnaire (RMDQ). The RMDQ is scored by adding up the number of items checked by the patient. The score can therefore range from 0 to 24. The original version of the Roland Morris Disability Questionnaire was published by Roland and Morris in 1983. A review of articles on the questionnaire was published in 2000 (Roland & Fairbank 2000). It comprises 24 items and measures the functional disability of patients with low back pain. This self-administered questionnaire is quick, easy to use, reliable, valid, and sensitive to changes in clinical status, suggesting that its use could be generalized in contexts ranging from epidemiological or clinical research to the individual assessment of patients with low back pain in everyday clinical practice. The questionnaire takes approximately 5 minutes to complete.
Functional disability in the experimental group (SM) | Month 3
  Functional disability will be measured according to the Roland Morris Disability Questionnaire (RMDQ). The RMDQ is scored by adding up the number of items checked by the patient. The score can therefore range from 0 to 24. The original version of the Roland Morris Disability Questionnaire was published by Roland and Morris in 1983. A review of articles on the questionnaire was published in 2000 (Roland & Fairbank 2000). It comprises 24 items and measures the functional disability of patients with low back pain. This self-administered questionnaire is quick, easy to use, reliable, valid, and sensitive to changes in clinical status, suggesting that its use could be generalized in contexts ranging from epidemiological or clinical research to the individual assessment of patients with low back pain in everyday clinical practice. The questionnaire takes approximately 5 minutes to complete.
Functional disability in the control group (PM) | Day 0
  Functional disability will be measured according to the Roland Morris Disability Questionnaire (RMDQ). The RMDQ is scored by adding up the number of items checked by the patient. The score can therefore range from 0 to 24. The original version of the Roland Morris Disability Questionnaire was published by Roland and Morris in 1983. A review of articles on the questionnaire was published in 2000 (Roland & Fairbank 2000). It comprises 24 items and measures the functional disability of patients with low back pain. This self-administered questionnaire is quick, easy to use, reliable, valid, and sensitive to changes in clinical status, suggesting that its use could be generalized in contexts ranging from epidemiological or clinical research to the individual assessment of patients with low back pain in everyday clinical practice. The questionnaire takes approximately 5 minutes to complete.
Functional disability in the control group (PM) | Month 1
  Functional disability will be measured according to the Roland Morris Disability Questionnaire (RMDQ). The RMDQ is scored by adding up the number of items checked by the patient. The score can therefore range from 0 to 24. The original version of the Roland Morris Disability Questionnaire was published by Roland and Morris in 1983. A review of articles on the questionnaire was published in 2000 (Roland & Fairbank 2000). It comprises 24 items and measures the functional disability of patients with low back pain. This self-administered questionnaire is quick, easy to use, reliable, valid, and sensitive to changes in clinical status, suggesting that its use could be generalized in contexts ranging from epidemiological or clinical research to the individual assessment of patients with low back pain in everyday clinical practice. The questionnaire takes approximately 5 minutes to complete.
Functional disability in the control group (PM) | Month 3
  Functional disability will be measured according to the Roland Morris Disability Questionnaire (RMDQ). The RMDQ is scored by adding up the number of items checked by the patient. The score can therefore range from 0 to 24. The original version of the Roland Morris Disability Questionnaire was published by Roland and Morris in 1983. A review of articles on the questionnaire was published in 2000 (Roland & Fairbank 2000). It comprises 24 items and measures the functional disability of patients with low back pain. This self-administered questionnaire is quick, easy to use, reliable, valid, and sensitive to changes in clinical status, suggesting that its use could be generalized in contexts ranging from epidemiological or clinical research to the individual assessment of patients with low back pain in everyday clinical practice. The questionnaire takes approximately 5 minutes to complete.
Pain management in the experimental group (SM) | In the week prior to inclusion
  The use of analgesics (Non-steroidal anti-inflammatory drugs, painkillers), lumbar braces, or osteopathic interventions will be recorded.
Pain management in the control group (PM) | In the week prior to inclusion
  The use of analgesics (Non-steroidal anti-inflammatory drugs, painkillers), lumbar braces, or osteopathic interventions will be recorded.
Pain management in the experimental group (SM) | Day 7 - 10 days
  The use of analgesics (Non-steroidal anti-inflammatory drugs, painkillers), lumbar braces, or osteopathic interventions will be recorded.
Pain management in the control group (PM) | Day 7 - 10 days
  The use of analgesics (Non-steroidal anti-inflammatory drugs, painkillers), lumbar braces, or osteopathic interventions will be recorded.
Pain management in the experimental group (SM) | Week 3
  The use of analgesics (Non-steroidal anti-inflammatory drugs, painkillers), lumbar braces, or osteopathic interventions will be recorded.
Pain management in the control group (PM) | Week 3
  The use of analgesics (Non-steroidal anti-inflammatory drugs, painkillers), lumbar braces, or osteopathic interventions will be recorded.
Pain management in the experimental group (SM) | Month 1
  The use of analgesics (Non-steroidal anti-inflammatory drugs, painkillers), lumbar braces, or osteopathic interventions will be recorded.
Pain management in the control group (PM) | Month 1
  The use of analgesics (Non-steroidal anti-inflammatory drugs, painkillers), lumbar braces, or osteopathic interventions will be recorded.
Pain management in the experimental group (SM) | Month 3
  The use of analgesics (Non-steroidal anti-inflammatory drugs, painkillers), lumbar braces, or osteopathic interventions will be recorded.
Pain management in the control group (PM) | Month 3
  The use of analgesics (Non-steroidal anti-inflammatory drugs, painkillers), lumbar braces, or osteopathic interventions will be recorded.
Need for a second consultation in the experimental group (SM) | Day 0 to Month 1
  The need for a second consultation with the manual physician within one month of the first consultation will be recorded
Need for a second consultation in the control group (PM) | Day 0 to Month 1
  The need for a second consultation with the manual physician within one month of the first consultation will be recorded
Number of medical visits in the experimental group (SM) | Day 7 - 10
  The number of medical visits made by the patient as part of their treatment for low back pain at each follow-up visit will be recorded
Number of medical visits in the control group (PM) | Day 7 - 10
  The number of medical visits made by the patient as part of their treatment for low back pain at each follow-up visit will be recorded
Number of medical visits in the experimental group (SM) | Month 1
  The number of medical visits made by the patient as part of their treatment for low back pain at each follow-up visit will be recorded
Number of medical visits in the control group (PM) | Month 1
  The number of medical visits made by the patient as part of their treatment for low back pain at each follow-up visit will be recorded
Number of medical visits in the experimental group (SM) | Month 3
  The number of medical visits made by the patient as part of their treatment for low back pain at each follow-up visit will be recorded
Number of medical visits in the control group (PM) | Month 3
  The number of medical visits made by the patient as part of their treatment for low back pain at each follow-up visit will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Nimes University Hospital, Nîmes, Gard, France